CLINICAL TRIAL: NCT04671719
Title: Autotaxin in Patients With GNAS/PTH Abnormalities
Brief Title: Determination of Circulating Autotaxin in Patients With GNAS or PTH Abnormalities
Acronym: GNAS-AUTAX
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0628
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Fibrous Dysplasia; Albright Syndrome; Adult Children; Hypoparathyroidism; Hyperparathyroidism; Pseudo Hypoparathyroidism
Keywords: Fibrous dysplasia / McCune-Albright syndrome, hypoparathyroidism, hyperparathyroidism, iPPSD, autotaxin, GNAS, PTH
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic; Hypoparathyroidism; Hyperparathyroidism; Pseudohypoparathyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sample — blood sample for circulating autotaxin measurement (5ml).

SUMMARY:
PTH secretion defects (grouped under the name hypoparathyroidism) are due to abnormalities in the PTH gene, abnormalities in the development of the parathyroid glands which synthesize PTH or abnormalities of the calcium sening receptor whose role is to adapt PTH level to ambient calcium level.

In contrast, primary hyperparathyroidism in children is also exceptional; expressed by hypercalcemia, with a renal and bon risk.

Pseudo-hypoparathyroidism, now known under the term inactivating PTH / PTHrP Signaling Disorder or iPPSD, are rare pathologies characterized by resistance to the action of PTH sometimes associated with other symptoms, in particular chondrodysplasia. They are linked to a defect in the action of a factor in the signaling pathway of G protein-coupled receptors that activate the production of cyclic AMP (cAMP). IPPSDs are most often due to a molecular defect in the GNAS gene, subject to parental imprint.

Fibrous dysplasia / McCune-Albright syndrome is a rare disease caused by somatic "gain-of-function" mutations in the GNAS gene located on chromosome 20q13 leading to activation of the protein Gαs and inappropriate production of intracellular cyclic adenosine monophosphate (cAMP). The clinical phenotype is determined by the location and extent of the tissues affected by this mutation.

Autotaxin (ATX) is a protein secreted by different tissues including the liver, fatty tissue, and bone. Today, ATX is described as the major source of LPA in the bloodstream. LPA interacts with one of its receptors on the surface of the cell membrane. Depending on the receptor engaged, one or more Gα subunits (G12 / 13, GQ, Gi / o or Gs) will activate multiple cell signaling pathways.

In bone, ATX is expressed by osteoclasts and osteoblasts. Recent laboratory data have shown that PTH stimulates ATX expression in osteoblasts in a dose-dependent manner.

The objective of this study is to provide clinical proof of concept that the PTH / Gαs / ATX pathway is truly significant in physiology and pathology, by studying the full spectrum of PTH and GNAS pathologies. If this proof of concept is obtained, therapeutic applications will probably be possible in the long term.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients :

* Children from 10 to 18 years old
* Patients with Fibrous dysplasia / McCune-Albright syndrome,hypoparathyroïdism, hyperparathyroïdism, or iPPSD, from References Centers for rare diseases (Calcium and phosphate metabolism, constitutional bone diseases) followed at hôpital Femme Mère Enfant (Bron) or at hôpital Bicêtre Paris Saclay (Paris).
* Patients and parent / holder of parental authority who have been informed of the study and do not object to participate

  • Adults:
* Patients > 18 years old
* Patients with Fibrous dysplasia / McCune-Albright syndrome, followed in reference center for constitutional bone diseases at hôpital Edouard Herriot (Lyon)
* Patients who have been informed of the study and do not object to participate

Exclusion Criteria:

* Children < 8 kg
* Patient with hepatic disease
* Patients under tutorship or curatorship
* Pregnant and / or breastfeeding woman
* Patient deprived of liberty
* Patient in emergency situation who can not agree to participate

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from 10 to 18 years old :
  1. Fibrous dysplasia / McCune-Albright syndrome,
  2. hypoparathyroïdism,
  3. hyperparathyroïdism,
  4. iPPSD, from References Centers for rare diseases (Calcium and phosphate metabolism, constitutional bone diseases) at hôpital Femme Mère Enfant (Bron) and at hôpital Bicêtre Paris Saclay (Paris).
  Adults with Fibrous dysplasia / McCune-Albright syndrome from reference center for constitutional bone diseases at hôpital Edouard Herriot (Lyon).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Concentration of circulating autotaxin | At inclusion
  Concentration of circulating autotaxin measured in patient serum by ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: BACCHETTA Justine, Pr, Principal Investigator — Centre de Référence des Maladies Rares du Calcium et du Phosphate
Locations (3):
- France (3):
  - Centre de compétence des maladies rares de l'insulino-sécrétion et de l'insulino-sensibilité, Bron
  - Centre de référence Dysplasie Fibreuse des os Service rhumatologie et pathologie osseuse Hôpital Edouard Herriot, Lyon, Lyon
  - Centre de Référence des Maladies Rares du Métabolisme du Calcium et du Phosphate Service d'Endocrinologie et Diabète de l'Enfant Hôpital Bicêtre Paris Saclay, Paris

IPD SHARING:
Plan to Share IPD: Undecided